CLINICAL TRIAL: NCT03569241
Title: PEACE V: a Randomized Phase II Trial for the Salvage Treatment of OligoRecurrent Nodal Prostate Cancer Metastases (STORM)
Brief Title: PEACE V: Salvage Treatment of OligoRecurrent Nodal Prostate Cancer Metastases
Acronym: STORM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2018/0130
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Metastatic Cancer; Oligometastatic Cancer
Keywords: Radiotherapy; metastasis-directed therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDT + ADT (Other): Metastasis-directed therapy (salvage lymph node dissection OR stereotactic body radiotherapy) + 6 months androgen deprivation therapy
  Interventions: Radiation: metastasis-directed treatment; Procedure: salvage Lymph Node Dissection; Drug: androgen deprivation therapy
- MDT + WPRT + ADT (Experimental): Metastasis-directed therapy (salvage lymph node dissection OR stereotactic body radiotherapy) + whole pelvic radiotherapy + 6 months androgen deprivation therapy
  Interventions: Radiation: whole pelvic radiotherapy; Radiation: metastasis-directed treatment; Procedure: salvage Lymph Node Dissection; Drug: androgen deprivation therapy

INTERVENTIONS:
Radiation: whole pelvic radiotherapy — addition of prophylactic whole pelvic radiotherapy to a local metastasis-directed treatment
  Arms: MDT + WPRT + ADT
Radiation: metastasis-directed treatment — stereotactic body radiotherapy
Procedure: salvage Lymph Node Dissection — metastasis-directed treatment
Drug: androgen deprivation therapy — LHRH-agonist (+ anti-androgen) or antagonist for a duration of 6 months

SUMMARY:
A proportion of prostate cancer (PCa) patients develop relapse following curative local treatment. Regional nodal recurrence is an emerging clinical situation since the introduction of new molecular imaging methods in the restaging of recurrent prostate cancer. More specifically, a subgroup of these patients is being diagnosed with a recurrence confined to the regional lymph nodes and limited in number (oligorecurrence) using choline or PSMA PET-CT. As there are no specific treatment recommendations for these type of patients, different treatment approaches are currently used, mostly focusing on local ablative treatments using radiotherapy or surgery. These treatments are coined metastasisdirected therapy (MDT). MDT in combination with or without temporary ADT could delay the subsequent risk of progression, and even cure limited regional nodal recurrences. Consequently, lifelong palliative ADT, with its toxicity and excess in non-cancer mortality might be postponed.

The proposed trial randomizes patients with oligorecurrent nodal prostate cancer following primary PCa treatment to either metastasis-directed therapy (MDT) (salvage lymph node dissection, sLND or stereotactic body radiotherapy, SBRT) or MDT plus whole pelvis radiotherapy (WPRT: 45 Gy in 25 fractions).

DETAILED DESCRIPTION:
A proportion of prostate cancer (PCa) patients develop a local, regional (N1) or distant (M1) relapse following curative local treatment. For both local and distant relapses, different treatment recommendations are made in the guidelines (EAU guidelines 2016). However, the entity regional nodal recurrence is not mentioned in the guidelines but is an emerging clinical situation since the introduction of choline and more recently PSMA PET-CT in the restaging of recurrent prostate cancer. More specifically, a subgroup of these patients is being diagnosed with a recurrence confined to the regional lymph nodes and limited in number (oligorecurrence) using choline or PSMA PET-CT. As there are no specific treatment recommendations for these type of patients, different treatment approaches are currently used, mostly focusing on local ablative treatments using radiotherapy or surgery. These treatments are coined metastasisdirected therapy (MDT). MDT in combination with or without temporary ADT could delay the subsequent risk of metastases, and even cure limited regional nodal recurrences. Consequently, lifelong palliative ADT, with its toxicity and excess in non-cancer mortality might be postponed.

The proposed trial randomizes patients with oligorecurrent nodal prostate cancer following primary PCa treatment to either metastasis-directed therapy (MDT) (sLND or SBRT) or MDT plus WPRT. In the recurrent PCa setting, 2 recent trials have suggested a progression-free and even survival benefit of adding temporary ADT to local salvage prostate bed radiotherapy. Consequently, this positive effect might also be applicable for regional recurrences. Although the optimal duration of ADT is unknown, a minimal duration of 6 months of ADT seems advisable in this setting and will be mandatory for both arms.

This trial will improve our insights in the pattern of recurrence following these treatment modalities with the expectation that WPRT will reduce the number of nodal relapses, improving metastasis-free survival and postponing the need for palliative systemic treatments while maintaining quality-of-life. The current phase II trial will try to establish a golden standard in the treatment of oligorecurrent nodal PCa.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of adenocarcinoma of the prostate
* Biochemical relapse of prostate cancer following radical local prostate treatment (radical prostatectomy, primary radiotherapy or radical prostatectomy +/- prostate bed adjuvant/ salvage radiotherapy) according to the EAU guidelines 2016.
* Following radical prostatectomy, patients with a biochemical relapse are eligible in case a nodal relapse is detected in the pelvis even in the absence of prior postoperative prostate bed radiotherapy (adjuvant or salvage).
* In case of a suspected local recurrence following primary radiotherapy, a biopsy should confirm local recurrence and patients with a confirmed local recurrence are eligible in case they also undergo a local salvage therapy. If imaging rules out local relapse, patients are eligible.
* Nodal relapse in the pelvis on choline, PSMA or FACBC PET-CT with a maximum of 3 positive nodal lymph nodes. The upper limit of the pelvis is defined as the aortic bifurcation.
* WHO performance state 0-1
* Age >18 years
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Bone or visceral metastases
* Para-aortic lymph node metastases (above the aortic bifurcation)
* Local relapse in the prostate gland or prostate bed not suitable for a curative treatment
* Previous irradiation of the pelvic and or para-aortic nodes
* Serum testosterone level <50ng/dl or 1.7 nmol/L at time of randomization
* Symptomatic metastases
* Lymph node metastases in previously irradiated areas resulting in dose constraint violation
* Contraindications to pelvic radiotherapy (chronic pelvic inflammatory bowel disease)
* Contraindications to androgen deprivation therapy
* PSA rise while on active treatment with (LHRH-agonist, LHRH-antagonist, anti-androgen, estrogen
* Previous treatment with cytotoxic agent for PCa
* Treatment during the past month with products known to influence PSA levels (e.g. fluconazole, finasteride, corticosteroids,…)
* Other active malignancy, except non-melanoma skin cancer or other malignancies with a documented disease-free survival for a minimum of 3 years before randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Metastases-free survival | 2 year
  Metastasis-free survival will be defined as the time between randomization and the appearance of a metastatic recurrence (any M1) as suggested by choline, FACBC or PSMA PET-CT or death due to any cause

SECONDARY OUTCOMES:
Clinical Progression free survival | 2 year
  Clinical Progression-free survival is defined as time between randomization and the appearance of a new recurrence (any N1 or M1) as suggested by PET-CT, symptoms related to progressive PCa, or death due to any cause
Biochemical progression-free survival | 2 year
  For patients who had previous RP at initial diagnosis, a biochemical recurrence is defined by any confirmed PSA rise above 0.20 ng/ml with a confirmatory rise at least 2 weeks later. For patients who had previous RT to the prostate at initial diagnosis, a biochemical recurrence is defined as the nadir + 2ng/ml (Phoenix definition). Non-responders are considered to have a biochemical recurrence in case a second measurement at least 2 weeks later confirms a rising PSA
Toxicity: acute toxicity | 3 months
  Radiotherapy toxicity will be assessed according to NCI CTCAE v4.0.
Toxicity: late toxicity | 2 year
  Radiotherapy toxicity will be assessed according to NCI CTCAE v4.0.
Patient reported QOL as per EORTC-QLQ C30 | 2 year
  Validated questionnaire assessing different health-related parameters (psychological, physical and social well-being) in cancer patients
Patient reported QOL as per EORTC-QLQ PR25 | 2 year
  Validated questionnaire assessing the health-related QOL of prostate cancer patients
Prostate cancer-specific survival | 5 year
  Cancer specific survival will be read as the time from trial randomization to the date of death due to prostate cancer
Overall survival | 5 year
  Overall survival will be read as the time from trial randomization to the date of death from any cause
Time to start of hormonal treatment | 2 year
  Time to hormonal treatment is defined as the time from trial randomization to start of hormonal treatment
Time to castration-resistant disease | 5 year
  Time to castration resistant disease is defined as the time from trial randomization until castration resistant status
economical evaluation | 2 year
  Assessment of quality-adjusted-life-years with the EuroQol classification system (EQ-5D-5L)
Sensitivity/specificity of PET-CT for the detection of nodal recurrences: limited to patients undergoing surgery | 3 months
  Sensitivity/specificity of PET-CT

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, PhD, Principal Investigator — University Hospital, Ghent
Locations (29):
- Epworth Healthcare, Melbourne, Australia
- Belgium (9):
  - GZA, Antwerp
  - AZ St-Jan Brugge, Bruges
  - AZ St-Lucas, Bruges
  - Institut Jules Bordet, Brussels
  - University Hospital Ghent, Ghent
  - AZ Maria Middelares, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CH Mouscron, Mouscron
- Italy (5):
  - Humanitas Research Hospital, Milan
  - Vita-Salute San Raffaele University, Milan
  - Istituto Nazionale Tumori IRCCS, Napoli
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Ospedale Sacro Cuore-Don Calabria, Verona
- Oslo University Hospital, Oslo, Norway
- Spain (8):
  - Cruces University Hospital, Barakaldo
  - Clínica Universitaria IMQ, Bilbao
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Universitario Quironsalud, Madrid
  - Hospitalario de Navarra, Navarro
  - Hospital Clínico de Santiago, Santiago
  - Hospital Universitari i Politècnic la Fe, Valencia
- Switzerland (5):
  - Universitätsspital Basel, Basel
  - Universitätsklinik für Radio-Onkologie, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ost P, Siva S, Brabrand S, Dirix P, Liefhooghe N, Otte FX, Gomez-Iturriaga A, Everaerts W, Shelan M, Conde-Moreno A, Lopez Campos F, Papachristofilou A, Guckenberger M, Scorsetti M, Zapatero A, Villafranca Iturre AE, Eito C, Counago F, Muto P, Duthoy W, Mach N, Fonteyne V, Moon D, Thon K, Mercier C, Achard V, Stellamans K, Goetghebeur E, Reynders D, Zilli T. Salvage metastasis-directed therapy versus elective nodal radiotherapy for oligorecurrent nodal prostate cancer metastases (PEACE V-STORM): a phase 2, open-label, randomised controlled trial. Lancet Oncol. 2025 Jun;26(6):695-706. doi: 10.1016/S1470-2045(25)00197-4. Epub 2025 May 5. PMID 40339593
- [Derived] Ost P, Siva S, Brabrand S, Dirix P, Liefhooghe N, Otte FX, Gomez-Iturriaga A, Everaerts W, Shelan M, Conde-Moreno A, Lopez Campos F, Papachristofilou A, Guckenberger M, Scorsetti M, Zapatero A, Villafranca Iturre AE, Eito C, Counago F, Muto P, Van De Voorde L, Mach N, Bultijnck R, Fonteyne V, Moon D, Thon K, Mercier C, Achard V, Stellamans K, Goetghebeur E, Reynders D, Zilli T. PEACE V-Salvage Treatment of OligoRecurrent nodal prostate cancer Metastases (STORM): Acute Toxicity of a Randomized Phase 2 Trial. Eur Urol Oncol. 2024 Jun;7(3):462-468. doi: 10.1016/j.euo.2023.09.007. Epub 2023 Oct 9. PMID 37821242
- [Derived] Huck C, Achard V, Zilli T. Surgical Treatments of Benign Prostatic Hyperplasia and Prostate Cancer Stereotactic Radiotherapy: Impact on Long-Term Genitourinary Toxicity. Clin Oncol (R Coll Radiol). 2022 Sep;34(9):e392-e399. doi: 10.1016/j.clon.2022.05.021. Epub 2022 Jun 15. PMID 35715340
- [Derived] Corkum MT, Achard V, Morton G, Zilli T. Ultrahypofractionated Radiotherapy for Localised Prostate Cancer: How Far Can We Go? Clin Oncol (R Coll Radiol). 2022 May;34(5):340-349. doi: 10.1016/j.clon.2021.12.006. Epub 2021 Dec 25. PMID 34961659
- [Derived] Zilli T, Dirix P, Heikkila R, Liefhooghe N, Siva S, Gomez-Iturriaga A, Everaerts W, Otte F, Shelan M, Mercier C, Achard V, Thon K, Stellamans K, Moon D, Conde-Moreno A, Papachristofilou A, Scorsetti M, Guckenberger M, Ameye F, Zapatero A, Van De Voorde L, Lopez Campos F, Counago F, Jaccard M, Spiessens A, Semac I, Vanhoutte F, Goetghebeur E, Reynders D, Ost P. The Multicenter, Randomized, Phase 2 PEACE V-STORM Trial: Defining the Best Salvage Treatment for Oligorecurrent Nodal Prostate Cancer Metastases. Eur Urol Focus. 2021 Mar;7(2):241-244. doi: 10.1016/j.euf.2020.12.010. Epub 2020 Dec 29. PMID 33386290
- [Derived] De Bruycker A, Spiessens A, Dirix P, Koutsouvelis N, Semac I, Liefhooghe N, Gomez-Iturriaga A, Everaerts W, Otte F, Papachristofilou A, Scorsetti M, Shelan M, Siva S, Ameye F, Guckenberger M, Heikkila R, Putora PM, Zapatero A, Conde-Moreno A, Counago F, Vanhoutte F, Goetghebeur E, Reynders D, Zilli T, Ost P. PEACE V - Salvage Treatment of OligoRecurrent nodal prostate cancer Metastases (STORM): a study protocol for a randomized controlled phase II trial. BMC Cancer. 2020 May 12;20(1):406. doi: 10.1186/s12885-020-06911-4. PMID 32398040